CLINICAL TRIAL: NCT04539236
Title: A Multicenter, Phase Ib/II Study That Combines Luspatercept and Lenalidomide (L2) in Lower-risk, Non-del(5q) MDS Patients
Brief Title: Luspatercept and Lenalidomide (L2) in Lower-risk, Non-del(5q) MDS Patients
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding Sponsor decision
Sponsor: Mikkael Sekeres, MD (Other)
Collaborators: Celgene (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Mikkael Sekeres, MD, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20201503; CASE2920 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: non-del(5q) MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide; luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Luspatercept + Lenalidomide Group (Experimental): Phase 1B: Luspatercept will be administered at starting dose 1.0 mg/kg and can be titrated to 1.33 and 1.75 mg/kg dependent on participant response. Lenalidomide will be administered in a dose escalation design between 3 cohorts to determine MTD (2.5 mg, 5 mg and 10 mg daily dose on a 21-day cycle). MTD will be defined as the dose level with 0 or 1 DLT out of 6 participants. MTD will be declared as the RP2D for the Phase II portion of the study.
  Phase II: Luspatercept will be administered at 1.0 mg/kg and can be titrated to 1.33 and 1.75 mg/kg dependent on participant response. Lenalidomide will be administered with the RP2D daily for 21 days on a 21 day cycle.
  Treatment with combination of Lenalidomide and Luspatercept will continue as long as a participant is deriving clinical benefit, in the opinion of the treating physician, for up to 5 years or until disease progression or treatment intolerance.
  Interventions: Drug: Lenalidomide; Drug: Luspatercept

INTERVENTIONS:
Drug: Lenalidomide — Administered daily by mouth on a 21 day cycle. Doses will be administered at 2.5 mg, 5 mg and 10 mg.
  Other Names: Revlimid
Drug: Luspatercept — Administered subcutaneously in the upper arm, thigh and/or abdomen on Day 1 of a 21 day cycle. Starting dose will be at 1.0 mg/kg and can be titrated, dependent on participant response, to doses of 1.33 mg/kg, and 1.75 mg/kg.
  Other Names: Reblozyl; ActRIIB-IgG; ACE-536; 1373715-00-4

SUMMARY:
The purpose of this study is to evaluate if the combination of drugs, Lenalidomide and Luspatercept, will help improve the treatment of anemia in patients with lower-risk Myelodysplastic Syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Documented diagnosis of MDS according to World Health Organization (WHO) / French-American-British (FAB) classification that meets International Prognostic Scoring System Revised (IPSS-R) classification (Greenberg, 2012) of very low, low, or intermediate risk disease; intermediate patients must have a blast percentage <5% to be enrolled.
4. Subjects can be ESA-naïve, or refractory or intolerant to, or ineligible for, prior ESA treatment, as defined by any one of the following:

   * Refractory to prior ESA treatment - documentation of non-response or response that is no longer maintained to prior ESA-containing regimen, either as single agent or combination (eg, with G-CSF); ESA regimen must have been either:

     * recombinant human erythropoietin (rHu EPO) ≥ 40,000 IU/wk for at least 8 doses or equivalent; OR
     * darbepoetin alpha ≥ 200-500 μg Q1-3W for at least 4 doses or equivalent;
   * Intolerant to prior ESA treatment - documentation of discontinuation of prior ESAcontaining regimen, either as single agent or combination (eg, with G-CSF), at any time after introduction due to intolerance or an adverse event
   * ESA ineligible - Low chance of response to ESA based on endogenous serum erythropoietin level > 200 U/L for subjects not previously treated with ESAs
5. If previously treated with ESAs, agents must have been discontinued ≥ 4 weeks prior to date of C1D1.
6. Requires RBC transfusions, as documented by the following criteria:

   * average transfusion requirement of ≥ 2 units/8 weeks of packed Red Blood Cells (pRBC)s preceding C1D1.
   * Hemoglobin levels at the time of or within 7 days prior to administration of a RBC transfusion must have been ≤ 10.0 g/dL for the transfusion to be counted towards meeting eligibility criteria. Red blood cell transfusions administered when Hgb levels were > 10.0 g/dL and/or RBC transfusions administered for elective surgery will not qualify as a required transfusion for the purpose of meeting eligibility criteria.
7. Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2 (Appendix 1)
8. Females of childbearing potential (FCBP), defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months), must:

   * Have two negative pregnancy tests (urine or serum) as verified by the Investigator prior to starting study therapy (unless the screening pregnancy test was done within 72 hours of C1D1). She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment.
   * If sexually active, agree to use, and be able to comply with, highly effective contraception without interruption, 5 weeks prior to starting investigational product, during the study therapy (including dose interruptions), and for 12 weeks after discontinuation of study therapy.
9. Male subjects must:

   * Agree to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (for example, polyurethane), during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 12 weeks following investigational product discontinuation, even if he has undergone a successful vasectomy.
10. Subject must have a negative Coronavirus Disease of 2019 (COVID-19) test completed ≤7 days prior to administration of protocol therapy.
11. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Prior therapy with Lenalidomide.
2. Previously treated with either luspatercept (ACE-536) or sotatercept (ACE-011)
3. MDS associated with del 5q cytogenetic abnormality
4. Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding

   * iron deficiency to be determined by serum ferritin ≤ 15 μg/L and additional testing if clinically indicated (eg, calculated transferrin saturation [iron/total iron binding capacity ≤ 20%] or bone marrow aspirate stain for iron).
5. Prior allogeneic stem cell transplant
6. Known history of diagnosis of AML
7. Use of any of the following within 4 weeks prior to C1D1:

   * anticancer cytotoxic chemotherapeutic agent or treatment
   * other RBC hematopoietic growth factors (eg, Interleukin-3)
   * investigational drug or device, or approved therapy for investigational use. If the half-life of the previous investigational product is known, use within 5 times the half-life prior to C1D1 or within 5 weeks, whichever is longer is excluded.
8. Uncontrolled hypertension, defined as repeated elevations of diastolic blood pressure (DBP) ≥ 100 mmHg despite adequate treatment.
9. Prior history of malignancies, other than MDS, unless the subject has been free of the disease (including completion of any active or adjuvant treatment for prior malignancy) for ≥ 1 year. However, subjects with the following history/concurrent conditions involving in situ cancer (or similar) are allowed:

   * Basal or squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis (TNM) clinical staging system)
10. Major surgery within 4 weeks prior to C1D1. Subjects must have completely recovered from any previous surgery prior to C1D1
11. History of stroke, deep venous thrombosis (DVT), pulmonary or arterial embolism within 6 months prior to C1D1
12. Pregnant or breastfeeding females
13. Subject has any significant medical condition, laboratory abnormality, psychiatric illness, or is considered vulnerable by local regulations (eg, imprisoned or institutionalized) that, in the opinion of the Investigator, would prevent the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
MTD/RP2D of Luspatercept combined with Lenalidomide | Up to 15 weeks
  Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of Luspatercept combined with Lenalidomide (reported in mg/kg) from Phase Ib portion of study
DLT Rate for Phase Ib | Up to 15 weeks
  DLT rate is defined as the percentage of participants with Dose Limiting Toxicities (DLT) as evaluated by treating physician using the National Cancer Center (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. DLTs are non-hematologic events grade 3 or higher that are at least possibly related to the investigational product and do not resolve to grade 1 or lower within 21 days.
Percentage of participants with RBC-TI response | Up to 5 years
  Red Blood Cell Transfusion Independence (RBC-TI) response is defined as participants who are RBC transfusion free over any consecutive 56-day period
Toxicity Rate for Phase II | Up to 5 years
  Toxicity rate is defined as the percentage of participants with treatment emergent adverse events (TE-AEs) as evaluated by treating physician using the National Cancer Center (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Percentage of participants with relevant reduction in RBC transfusion requirement | Up to 5 years
  Participants with relevant reduction in RBC transfusion requirement will be defined as those participants whose total number of RBC units transfused has decreased by at least 4 units compared to the number transfused during the 8 weeks before study participation
Percentage of participants with Erythroid Response | Up to 5 years
  Hematologic Improvement Erythroid Response (HI-E) will bdefined as at least a 1.5 g/dl increase in serum hemoglobin from baseline
Duration of RBC-TI | Up to 5 years
  The length of time where participants are RBC transfusion free will be reported
Percentage of participants with Platelet Response | Up to 5 years
  Hematologic improvement Platelet response (HI-P) will be defined as:
  For participants with a serum baseline platelet count of > 20,000/mm3 at baseline: An absolute increase of ≥ 30,000/mm3 from baseline
  For participants with a serum platelet count ≤ 20,000/mm3 at baseline: An increase of at least 100% from baseline counts to a platelet count > 20,000/mm3.
Percentage of participants with Neutrophil Response | Up to 5 years
  Hematologic improvement of Neutrophil Response (HI-N) will be defined as a serum absolute neutrophil count (ANC) increase from baseline of at least 100%, and an absolute increase of > 500/mm3 from baseline.
Percentage of participants experiencing a progression to higher-risk MDS or AML | Up to 5 years
  Percentage of participants experiencing a progression to higher-risk Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML)
Overall Survival (OS) | Up to 5 years
  OS is calculated for all participants from the date of initial registration to date of death due to any cause. The follow-up for participants last known to be alive is censored at the date of last contact.
Percentage of participants with RBC-TI lasting 16 weeks | Up to 5 years
  Percentage of participants with RBC-TI lasting 16 weeks (112 days) will be assessed per the Blood 2019 position paper on defining response in lower-risk MDS

CONTACTS AND LOCATIONS:
Overall Officials: Mikkael Sekeres, MD, Principal Investigator — University of Miami
Locations (5):
- United States (5):
  - University of Miami, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No